CLINICAL TRIAL: NCT05778799
Title: Balance Assessment of People With Lower Limb Impairment Practicing Amputee Football
Brief Title: Physical Activity and Sports for People With Special Needs
Status: Completed | Type: Observational
Sponsor: Józef Piłsudski University of Physical Education (Other)
Responsible Party: Sponsor
Other Study IDs: Research Group no 4
Record Dates: First submitted 2023-03-10; First posted 2023-03-21 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Amputation; Dysmelia; Leg; Deformity, Congenital
Keywords: Amputation; Amputee Football; Performance; Balance
MeSH Terms: conditions — Lower Extremity Deformities, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Balance test — 10 second left- or right-leg stance with eyes open, and single 10 second left- or right-leg stance with eyes closed

SUMMARY:
Purpose of this study was to assess the balance level of highly qualified amputee football players in relation to their sports level, training experience, position on the pitch, as well as the type of amputation/dysfunction and disability experience.

DETAILED DESCRIPTION:
The participants were presented with the procedure of the study and informed that they could resign from their participation in the study at any stage. All participants were given the written informed consent form after the detailed written and oral explanation of the risk and benefits resulting from participation in this study Static balance was assessed using AMTI AccuSway stabilographic platform (ACS Model). The study participants performed the single 10 second left- or right-leg stance with eyes open (EO), and single 10 second left- or right-leg stance with eyes closed (EC) (depending on leg amputation). If the first attempt was not successful, study participants were able to do the second attempt. The tests were conducted on a match-free day, approximately 2 hours after a meal, in a sports outfit, in a specially designated room.

ELIGIBILITY:
Inclusion Criteria:

* participant of European Amputte Football Championschip
* field player (leg amputation or leg dysfunction)
* written consent form

Exclusion Criteria:

* goalkeeper
* injury
* tiredness
* refusal

Min Age: 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Members of 14 teams, field players with lower limb impairment participating in European Amputee Football Championship.
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2021-09-11 (Actual); Primary Completion 2021-09-19 (Actual); Study Completion 2021-09-19 (Actual)

PRIMARY OUTCOMES:
Center of pressure (CoP) path lenght was measured | Baseline
  CoP displacement analysis is used to assess postural sway, based on which the balance control function can be assessed
Surface area of stabilogram was mesured | Baseline
  Based on the analysis of the surface area of the stabilogram, the level of balance control can be assessed
Visual inspection indicator (VII) was measured | Baseline
  VII aggregates surface areas of stabilograms (cm2) with eyes open and closed. In theory, maximum value of the indicator may come to 100%. As a rule, it is positive, which means that the surface area of the stabilogram increases with eyes closed. The indicator is higher when the difference between the surface area of the stabilogram in the test with eyes closed and the surface area of the stabilogram in the test with eyes open is greater. Lower values of the VII may indicate a reduced role of visual control in maintaining balance or the lack of its compensation.

CONTACTS AND LOCATIONS:
Overall Officials: Jolanta Marszałek, PhD, Study Director — University of Physical Education in Warsaw
Locations (1):
- University of Physical Education, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Role of vision in static balance in persons with and without visual impairments — https://pubmed.ncbi.nlm.nih.gov/33541039/
- See also: Effects of sport on static balance in athletes with visual impairments — https://pubmed.ncbi.nlm.nih.gov/30421870/